CLINICAL TRIAL: NCT01996839
Title: Loteprednol Etabonate Ophthalmic Gel, 0.38% (BID and TID) Versus Vehicle Gel for the Treatment of Ocular Inflammation and Pain Following Cataract Surgery
Brief Title: Loteprednol Ophthalmic Gel for the Treatment of Ocular Inflammation and Pain Following Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 842
Record Dates: First submitted 2013-11-22; First posted 2013-11-27 (Estimated); Results first posted 2020-09-03 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Inflammation; Pain; Cataract
MeSH Terms: conditions — Inflammation; Pain; Cataract | interventions — BID protein, human; Loteprednol Etabonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Loteprednol Etabonate Gel (BID) (Experimental): Loteprednol Etabonate Gel 0.38% administered two times daily (BID).
  Interventions: Drug: Loteprednol Etabonate Gel (BID)
- Vehicle (BID) (Active Comparator): Vehicle of Loteprednol Etabonate Gel 0.38% administered two times daily (BID).
  Interventions: Drug: Vehicle (BID)
- Loteprednol Etabonate Gel (TID) (Experimental): Loteprednol Gel 0.38% administered three times daily (TID).
  Interventions: Drug: Loteprednol Etabonate Gel (TID)
- Vehicle (TID) (Active Comparator): Vehicle of Loteprednol Etabonate Gel 0.38% administered three times daily (TID).
  Interventions: Drug: Vehicle (TID)

INTERVENTIONS:
Drug: Loteprednol Etabonate Gel (BID) — One drop of LE gel instilled into the study eye two times per day (BID) for 14 days
  Other Names: Lotemax
  Arms: Loteprednol Etabonate Gel (BID)
Drug: Loteprednol Etabonate Gel (TID) — One drop of LE gel instilled into the study eye three times per day (TID) for 14 days.
  Other Names: Lotemax
  Arms: Loteprednol Etabonate Gel (TID)
Drug: Vehicle (BID) — One drop of vehicle instilled into the study eye two times per day (BID) for 14 days
  Other Names: Vehicle
  Arms: Vehicle (BID)
Drug: Vehicle (TID) — One drop of vehicle instilled into the study eye three times per day (TID) for 14 days
  Other Names: Vehicle
  Arms: Vehicle (TID)

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of loteprednol etabonate ophthalmic gel

DETAILED DESCRIPTION:
The objective of this study is to evaluate the safety and efficacy of loteprednol etabonate ophthalmic gel, 0.38% (BID and TID) for the treatment of postoperative inflammation and pain following cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

Visit 1 (Screening Visit)

* Be willing and able to comply with all treatment and follow-up/study procedures.
* Be a candidate for routine, uncomplicated cataract surgery

Visit 3 (Postoperative Day 1)

* Have undergone routine, uncomplicated cataract surgery (phaco- emulsification with posterior chamber IOL implantation, not combined with any other surgery) in the study eye.
* Have ≥ Grade 2 anterior chamber (AC) cells (6-15 cells) in the study eye.

Exclusion Criteria:

* Have a severe/serious ocular condition or history/presence of chronic generalized systemic disease that the Investigator feels might increase the risk to the subject or confound the result(s) of the study.
* Have known hypersensitivity or contraindication to the study drug(s) or their components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2013-12; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon I Williams, PhD, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb Incorporated, Bridgewater, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The 2 vehicle arms were combined into 1 treatment group in the statistical analysis, and hence the study has 3 treatment groups (ie, Loteprednol Etabonate Gel TID, Loteprednol Etabonate Gel BID, and [combined] vehicle groups).
Groups:
- Vehicle (BID and TID): Vehicle of Loteprednol Etabonate Gel 0.38% administered two times daily (BID) and three times daily (TID), combined arms
  One drop of vehicle instilled into the study eye two times per day (BID) and three times a day (TID) for 14 days
Period: Overall Study
Arm/Group | Vehicle (BID and TID) | Loteprednol Etabonate Gel (BID) | Loteprednol Etabonate Gel (TID)
Started | 172 | 171 | 171
Completed | 80 | 133 | 139
Not Completed | 92 | 38 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle (BID and TID) | Loteprednol Etabonate Gel (BID) | Loteprednol Etabonate Gel (TID) | Total
Number analyzed (Participants) | 172 | 171 | 171 | 514
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (8.56) | 70.0 (8.34) | 70.5 (8.15) | 69.8 (8.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 94 | 89 | 283
  Male | 72 | 77 | 82 | 231

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Resolution of Anterior Chamber (AC) Cells
Description: White blood cell accumulation in anterior aqueous humor was assessed by the Investigator during slit lamp examination and graded on a 5-point scale: Grade 0 = no cells seen; Grade 1 = 1 to 5 cells; Grade 2 = 6 to 15 cells; Grade 3 = 16 to 30 cells; Grade 4 = > 30 cells. Lower score indicated better outcome. Complete resolution of AC cells was defined as cell score = 0 in the study eye.
Time Frame: 8 days
Population: The analysis population included all randomized participants, with missing values imputed as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle (BID and TID) | Loteprednol Etabonate Gel (BID) | Loteprednol Etabonate Gel (TID)
Number analyzed (Participants) | 172 | 171 | 171
Participants | 16 | 46 | 49

2. Primary Outcome: Percentage of Participants With Grade 0 Pain in the Study Eye.
Description: Ocular pain, defined as a positive sensation of the eye, including foreign body sensation, stabbing, throbbing, or aching, was assessed and graded by subjects on the 6-point scale, with 0=None and 5=Severe.
Time Frame: 8 days
Population: The analysis population included all randomized participants, with missing values imputed as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle (BID and TID) | Loteprednol Etabonate Gel (BID) | Loteprednol Etabonate Gel (TID)
Number analyzed (Participants) | 172 | 171 | 171
Participants | 82 | 126 | 125

3. Secondary Outcome: Percentage of Participants With Complete Resolution of Anterior Chamber (AC) Cells by Visit
Description: as for outcome 1
Time Frame: 18 days
Population: The analysis population included all randomized participants, with missing values imputed as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle (BID and TID) | Loteprednol Etabonate Gel (BID) | Loteprednol Etabonate Gel (TID)
Number analyzed (Participants) | 172 | 171 | 171
Participants
  Day 3 | 12 | 13 | 7
  Day 15 | 28 | 73 | 83
  Day 18 | 40 | 77 | 91

4. Secondary Outcome: Percentage of Participants With Grade 0 Pain in the Study Eye by Visit.
Description: as for outcome 1
Time Frame: 18 days
Population: The analysis population included all randomized participants, with missing values imputed as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle (BID and TID) | Loteprednol Etabonate Gel (BID) | Loteprednol Etabonate Gel (TID)
Number analyzed (Participants) | 172 | 171 | 171
Participants
  Day 3 | 96 | 123 | 117
  Day 15 | 81 | 129 | 137
  Day 18 | 73 | 122 | 122

5. Secondary Outcome: Percentage of Participants With Complete Resolution of Anterior Chamber (AC) Flare in the Study Eye by Visit.
Description: Flare was evaluated by the Investigator by assessing the scattering of a slit lamp light beam directed into the anterior chamber (Tyndall effect). Flare was graded on the 5-point scale, with 0=None (best) and 4=Very Severe (worst). Complete resolution of AC flare was defined as Grade 0.
Time Frame: 18 days
Population: The analysis population included all randomized participants, with missing values imputed as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle (BID and TID) | Loteprednol Etabonate Gel (BID) | Loteprednol Etabonate Gel (TID)
Number analyzed (Participants) | 172 | 171 | 171
Participants
  Day 3 | 78 | 95 | 90
  Day 8 | 71 | 117 | 122
  Day 15 | 71 | 124 | 131
  Day 18 | 68 | 115 | 127

6. Secondary Outcome: Percentage of Participants With Complete Resolution of Anterior Chamber (AC) Cells and AC Flare in the Study Eye by Visit.
Description: White blood cell accumulation in anterior aqueous humor was assessed by the Investigator during slit lamp examination and graded on a 5-point scale: Grade 0 = no cells seen; Grade 1 = 1 to 5 cells; Grade 2 = 6 to 15 cells; Grade 3 = 16 to 30 cells; Grade 4 = > 30 cells. Lower score indicated better outcome. Complete resolution of AC cells was defined as cell score = 0 in the study eye. Flare was evaluated by the Investigator by assessing the scattering of a slit lamp light beam directed into the anterior chamber (Tyndall effect). Flare was graded on the 5-point scale, with 0=None (best) and 4=Very Severe (worst).
Time Frame: 18 days
Population: The analysis population included all randomized participants, with missing values imputed as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle (BID and TID) | Loteprednol Etabonate Gel (BID) | Loteprednol Etabonate Gel (TID)
Number analyzed (Participants) | 172 | 171 | 171
Participants
  Day 3 | 11 | 12 | 7
  Day 8 | 16 | 45 | 47
  Day 15 | 27 | 73 | 83
  Day 18 | 40 | 74 | 90

ADVERSE EVENTS:
Time Frame: 18 days
Description: The safety analysis population included all randomized participants who received treatment. There was one participant who did not receive treatment, thus there were 513 participants in the safety population.
Arm/Group | Vehicle (BID and TID) | Loteprednol Etabonate Gel (BID) | Loteprednol Etabonate Gel (TID)
All-Cause Mortality (participants affected / at risk) | 0/172 | 0/171 | 0/170
Serious Adverse Events (participants affected / at risk) | 1/172 | 1/171 | 0/170
Other Adverse Events (participants affected / at risk) | 0/172 | 0/171 | 0/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle (BID and TID) (N=172) | Loteprednol Etabonate Gel (BID) (N=171) | Loteprednol Etabonate Gel (TID) (N=170)
Endophthalmitis (Eye disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.